CLINICAL TRIAL: NCT01112163
Title: The Effect of Enhanced External Counter Pulsation on Left Ventricular Systolic and Diastolic Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Herning Hospital (Other)
Responsible Party: Medicinsk Afdeling Regionshospitalet Herning, Hospitalenheden Vest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EECP-VV
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-03

CONDITIONS: Ischemic Heart Disease
Keywords: ischemic heart disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced external counter pulsation (Experimental): One session of enhanced external counter pulsation (60 minutes)
  Interventions: Device: Enhanced external counter pulsation

INTERVENTIONS:
Device: Enhanced external counter pulsation — While an individual is undergoing ECP, they have pneumatic stockings (also known as cuffs) on their legs and are connected to telemetry monitors that monitor their heart rate and rhythm.The cuffs should ideally inflate at the beginning of diastole and deflate at the beginning of systole. During the inflation portion of the cycle, the calf cuffs inflate first, then the lower thigh cuffs and finally the upper thigh cuffs. Inflation is controlled by a pressure monitor, and the cuffs are inflated to about 300 mmHg.

SUMMARY:
Enhanced external counter pulsation (EECP) is a procedure performed on patients with ischemic heart disease. The treatment improves physical capacity and relieves angina pectoris. It is suitable for patients with persistent angina pectoris despite and for patients not amendable for coronary revascularization. Some studies demonstrate a relationship between diastolic and systolic blood pressure ratio (d/s ratio) and the effect of EECP.

The aim of the investigators study is to understand the effect of EECP on left ventricular systolic and diastolic function assessed by trans-thoracic echocardiography (TTE).

Hypothesis: EECP improves left ventricular systolic and diastolic function. There is a relationship between d/s ratio and aortic arterial stiffness EECP improves left ventricular diastolic function Standard TTE would be performed prior the EECP procedure, which lasts 60 min., and repeated every 15 minutes. Moreover the investigators would measure pulse wave velocity, a measure of aortic arterial stiffness, in order to investigate the relationship between the d/s ratio and arterial stiffness.

The patients would be recruited among former study patients who have undergone EECP before. 20 patients with the best acoustic conditions would be selected and invited to enroll into the study.

ELIGIBILITY:
Inclusion Criteria:

* Angina pectoris, CCS-class 2-4
* Reversal ischemia
* Pathological coronary angiogram without the possibility of revascularization
* Sinus rhythm

Exclusion Criteria:

* Cancer
* Dementia
* Pregnancy
* Blood pressure > 180/110
* Severe valvular disease
* Ejection fraction < 25%
* Acute coronary syndrome the last 3 months
* History of aortic aneurism
* Pacemaker
* Diabetes mellitus
* Cardiac arrythmia that prevents the EECP procedure
* Bleeding
* Active venous thrombosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricular longitudinal strain | 60 minutes
  A measure of left ventricular shortening during systole assessed by speckle tracking with trans thoracic echocardiography

SECONDARY OUTCOMES:
Pulse wave velocity | 60 minutes
  Pulse wave velocity is a measure of aortic arterial stiffness. The outcome is the relationhip between pulse wave velocity and d/s ratio
left ventricular diastolic function | 60 minutes
  EECP reduces left ventricular after load and increases cardiac output. Left ventricular diastolic function is assessed by tissue Doppler imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Eftekhari, MD PhD, Principal Investigator — Regionshospitalet Herning / Dept. Pharmacology Aarhus University; Ole May, MD PhD, Study Chair — Herning Hospital
Locations (1):
- Regionshospitalet Herning, Herning, Denmark

REFERENCES:
- [Derived] May O, Sogaard HJ. Enhanced External Counterpulsation Is an Effective Treatment for Depression in Patients With Refractory Angina Pectoris. Prim Care Companion CNS Disord. 2015 Aug 20;17(4):10.4088/PCC.14m01748. doi: 10.4088/PCC.14m01748. eCollection 2015. PMID 26693035